CLINICAL TRIAL: NCT05601791
Title: Efficacy of Percutaneous Laser Disc Decompression Versus Epidural Steroid and Local Anesthetic Injection by Transforaminal Approach in the Treatment of Lumbar Radicular Pain
Brief Title: Efficacy of PLDD Versus ESI in the Treatment of Lumbar Radicular Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Osijek University Hospital (Other)
Responsible Party: Principal Investigator, Dino Budrovac, MD, Specialist in anesthesiology, resuscitation and intensive care medicine, Osijek University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2158-61-07-20-05
Record Dates: First submitted 2022-10-12; First posted 2022-11-01 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Herniated Disc; Low Back Pain
Keywords: herniated disc; epidural injection; laser; low back pain; radiculopathy
MeSH Terms: conditions — Intervertebral Disc Displacement; Low Back Pain; Radiculopathy

STUDY DESIGN:
Intervention Model Description: The research is designed as a randomized controlled trial, and will be conducted at the Clinic for Anesthesiology, Reanimatology and Intensive Medicine in the Department of Pain Management of the Osijek Clinical Hospital Center after obtaining the approval of the Ethics Committee. All patients will receive a written informed consent in which the procedure to be performed will be described, and the procedure will also be explained to them orally. After signing the informed consent, the patients will be divided into 2 groups using a random number generator, depending on whether there is discorradicular contact or not, and then according to the treatment method (ESI TF or PLDD). All subjects will be selected at the Institute for Pain Management of KBC Osijek.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Discoradicular contact+ESI TF (Active Comparator): Patients with discorradicular contact who underwent ESI TF
  Interventions: Procedure: Epidural Steroid Injection
- Discoradicular contact+PLDD (Active Comparator): Patients with discorradicular contact who underwent PLDD
  Interventions: Procedure: Percutaneous Laser Disc Decompression
- Without discoradicular contact+ESI TF (Active Comparator): Patients without discorradicular contact who underwent ESI TF
  Interventions: Procedure: Epidural Steroid Injection
- Without discoradicular contact+PLDD (Active Comparator): Patients without discorradicular contact who underwent PLDD
  Interventions: Procedure: Percutaneous Laser Disc Decompression

INTERVENTIONS:
Procedure: Epidural Steroid Injection — Epidural Steroid Injection transforaminal approach Drug: midazolam, fentanyl, lidocaine, levobupivacaine, methilprednisoloneacetat
  Arms: Discoradicular contact+ESI TF; Without discoradicular contact+ESI TF
Procedure: Percutaneous Laser Disc Decompression — Percutaneous Laser Disc Decompression Drug: midazolam, fentanyl, lidocaine
  Arms: Discoradicular contact+PLDD; Without discoradicular contact+PLDD

SUMMARY:
The most common cause of lumbar radicular pain is intervertebral disc herniation with or without pressure on the nerve root, which leads to inflammation and pain. Just as the mechanical component is important, so is the inflammatory component in the etiology of lumbar radicular pain. Numerous pro-inflammatory and anti-inflammatory proteins were found in serum, cerebrospinal fluid and disc biopsies from patients with lumbar radicular pain. Interleukin(IL)-1β, IL-6, IL-8, and tumor necrosis factor TNF-α are the most frequently investigated (8, 9).

Elevated levels of IL-6 and TNF-α were found in patients with lumbar pain caused by intervertebral disc herniation.

In order to avoid systemic and unwanted effects of analgesics, undergoing anesthesia and long-term and extensive operations, minimally invasive procedures are increasingly used in the treatment of lumbar radicular pain. Epidural administration of steroids and local anesthetic through a transforaminal approach (ESI TF) and percutaneous laser disc decompression (PLDD) are some of these methods.

Lumbar radicular pain occurs due to inflammation and/or disc-radicular contact. Corticosteroids interrupt the inflammatory process, the transmission of pain signals via nociceptive C fibers and reduce capillary permeability. Along with the corticosteroid, a local anesthetic is also applied, which leads to immediate analgesia by blocking the conduction of painful impulses by blocking sodium channels. Percutaneous laser disc decompression (PLDD) is a minimally invasive method of treating lumbar radicular pain performed under local anesthesia under fluoroscopic control. The laser energy leads to the heating of the tissue of the nucleus pulposus, which leads to the evaporation of a small volume of water inside the disc. Viewing the disc as a closed hydraulic system, a small decrease in the water content within the disc leads to a disproportionate decrease in intradiscal pressure, which results in retraction of the herniated disc. Thermal energy leads to protein denaturation, which causes structural changes and thus prevents further retention of water in the disc, and a stable scar is created at the point of laser action. On the basis of current knowledge, an attempt is made to establish a link between inflammatory parameters as predictive and prognostic biomarkers in the treatment of patients with lumbar radicular pain caused by intervertebral disc herniation.

DETAILED DESCRIPTION:
The hypothesis is that:

* there will be no difference in effectiveness in reducing the intensity of pain, improving the quality of life, reducing the degree of disability, reducing neuropathic pain, reducing anxiety and depression, and improving the quality of sleep in the treatment of lumbar radicular pain caused by disc herniation without discoradicular contact, but PLDD will be more effective in patients where there is discorradicular contact
* PLDD will lead to a greater reduction in serum levels of inflammatory markers in patients with nerve compression by intervertebral disc herniation
* ESI TF will lead to a greater reduced serum level of inflammatory markers where there is no nerve compression by intervertebral disc herniation
* The group of patients in whom PLDD was performed will have a significantly greater retraction of the disc herniation compared to ESI TF

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 60
* Signing informed consent
* Unilateral lumbar radicular pain
* Subjects who do not responds to conservative treatment
* Disc herniation at one level
* MR verified disc herniation
* Pain intensity measured by VAS scale, from 0 - 10, >5

Exclusion Criteria:

* Subjects younger than 18 and older than 65 years
* Refusal of the subjects to participate in the research
* Central stenosis of the lumbar canal
* Lumbar radicular pain caused by causes other than intervertebral disc herniation
* Pregnancy
* Allergy to steroids, local anesthetics, fentanyl, midazolam and contrast medium
* Positive history of prolonged bleeding
* Local or systemic infection
* Previous lumbar spine surgery7
* Opioid abuse
* Proven inflammatory rheumatic disease and inflammatory bowel disease in the active phase
* Other acute infections

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Compare the effectiveness in reducing pain intensity with ESI TF and PLDD in patients with lumbar radicular pain caused by intervertebral disc herniation | Six months
  Compare the effectiveness in reducing pain intensity with epidural administration of steroids and local anesthetic through a transforaminal approach (ESI TF) and percutaneous laser disc decompression (PLDD) in patients with lumbar radicular pain caused by intervertebral disc herniation, measured by the VAS scale (0-10). The severity of pain was assessed using the visual-analog scale of pain (VAS). The scale consists of a solid line that is 0 to 10 numbered at both its beginning and conclusion. The number 0, which denotes the lack of pain, is located on the far left, while the number 10, which denotes unbearable pain, is located on the far right.
Investigate the difference imeasured with a visual analogue scale between ESI TF and PLDD in herniated intervertebral disc with and without discoradicular contact | Six months
  Investigate the difference measured with a visual analogue scale between ESI TF and PLDD in herniated intervertebral disc with and without discoradicular contact. The severity of pain was assessed using the visual-analog scale of pain (VAS). The scale consists of a solid line that is 0 to 10 numbered at both its beginning and conclusion. The number 0, which denotes the lack of pain, is located on the far left, while the number 10, which denotes unbearable pain, is located on the far right.

SECONDARY OUTCOMES:
Investigate the influence of ESI TF and PLDD on the serum level of interleukin-6 (IL-6) | Six months
  Investigate the influence of ESI TF and PLDD on the serum level of interleukin-6 (IL-6)
Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on quality of life | Six months
  Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on quality of life measured by SF-36 (Short form health survey-36). The Health Status Questionnaire SF-36 was used to examine health status and health-related quality of life. The questionnaire is intended for self-assessment of mental and physical health and social functioning. The SF-36 is a short health status questionnaire consisting of 36 questions. The score is expressed as a standardized value ranging from 0 to 100 for each dimension. Low scores reflect reduced and limited functionality, i.e. loss of function, existence of pain and poor health assessment. High scores reflect the assessment of health as good, without pain and without functional limitations.
Investigate the influence of PLDD and ESI TF on the retraction of disc herniation | Six months
  Investigate the influence of PLDD and ESI TF on the retraction of disc herniation which will be measured by MR control after 6 months
Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on degree of disability | Six months
  Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on degree of disability measured by Oswestry Disability Questionnaire Index (ODI). The degree of disability for carrying out everyday activities as a result of low back pain will be evaluated using the Oswestry Disability Index (ODI) questionnaire. The domains of the questionnaire cover aspects of pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sexual function, social life, and traveling, each one containing six statements about section-related activities. The responses are scored on a 0-5 scale. Total score is expressed as the percentage of the maximum score with lower scores indicating lower levels of disability and vice versa.
Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on neuropathic pain | Six months
  Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on neuropathic pain measured by Pain Detect. The Pain Detect questionnaire is a standardized questionnaire for screening the probability of the existence of a neuropathic pain component in patients with chronic pain. It consists of three parts in sequence from the assessment of the intensity of the pain through the pictorial presentation of the nature of the pain and the main area of the pain to the final questions about the severity of the sensory symptoms which are classified into five groups according to the intensity, from never to very severe.
Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on degree of anxiety and depression | Six months
  Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on degree of anxiety and depression measured by the Hospital Anxiety and Depression Scale (HADS). The HADS questionnaire has seven items each for depression and anxiety subscales. Scoring for each item ranges from zero to three, with three denoting highest anxiety or depression level. A total subscale score of >8 points out of a possible 21 denotes considerable symptoms of anxiety or depression.
Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on quality of sleep | Six months
  Investigate the impact of PLDD and ESI TF in the treatment of lumbar radicular pain caused by disc herniation on quality of sleep measured by the Pittsburgh Sleep Quality Index (PSQI), consisting of 19 items, each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Dino Budrovac, MD, Principal Investigator — UH Osijek
Locations (1):
- UH Osijek, Osijek, Croatia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hoy D, March L, Brooks P, Blyth F, Woolf A, Bain C, Williams G, Smith E, Vos T, Barendregt J, Murray C, Burstein R, Buchbinder R. The global burden of low back pain: estimates from the Global Burden of Disease 2010 study. Ann Rheum Dis. 2014 Jun;73(6):968-74. doi: 10.1136/annrheumdis-2013-204428. Epub 2014 Mar 24. PMID 24665116
- [Background] Khan AN, Jacobsen HE, Khan J, Filippi CG, Levine M, Lehman RA Jr, Riew KD, Lenke LG, Chahine NO. Inflammatory biomarkers of low back pain and disc degeneration: a review. Ann N Y Acad Sci. 2017 Dec;1410(1):68-84. doi: 10.1111/nyas.13551. PMID 29265416
- [Background] Porchet F, Wietlisbach V, Burnand B, Daeppen K, Villemure JG, Vader JP. Relationship between severity of lumbar disc disease and disability scores in sciatica patients. Neurosurgery. 2002 Jun;50(6):1253-9; discussion 1259-60. doi: 10.1097/00006123-200206000-00014. PMID 12015843
- [Background] el Barzouhi A, Vleggeert-Lankamp CL, Lycklama a Nijeholt GJ, Van der Kallen BF, van den Hout WB, Jacobs WC, Koes BW, Peul WC; Leiden-The Hague Spine Intervention Prognostic Study Group. Magnetic resonance imaging in follow-up assessment of sciatica. N Engl J Med. 2013 Mar 14;368(11):999-1007. doi: 10.1056/NEJMoa1209250. PMID 23484826
- [Background] Wuertz K, Haglund L. Inflammatory mediators in intervertebral disk degeneration and discogenic pain. Global Spine J. 2013 Jun;3(3):175-84. doi: 10.1055/s-0033-1347299. Epub 2013 May 21. PMID 24436868
- [Background] Jungen MJ, Ter Meulen BC, van Osch T, Weinstein HC, Ostelo RWJG. Inflammatory biomarkers in patients with sciatica: a systematic review. BMC Musculoskelet Disord. 2019 Apr 9;20(1):156. doi: 10.1186/s12891-019-2541-0. PMID 30967132
- [Background] Kraychete DC, Sakata RK, Issy AM, Bacellar O, Santos-Jesus R, Carvalho EM. Serum cytokine levels in patients with chronic low back pain due to herniated disc: analytical cross-sectional study. Sao Paulo Med J. 2010;128(5):259-62. doi: 10.1590/s1516-31802010000500003. PMID 21181064
- [Background] Patel VB, Wasserman R, Imani F. Interventional Therapies for Chronic Low Back Pain: A Focused Review (Efficacy and Outcomes). Anesth Pain Med. 2015 Aug 22;5(4):e29716. doi: 10.5812/aapm.29716. eCollection 2015 Aug. PMID 26484298
- [Background] Harris JD. Management of expected and unexpected opioid-related side effects. Clin J Pain. 2008 May;24 Suppl 10:S8-S13. doi: 10.1097/AJP.0b013e31816b58eb. PMID 18418226
- [Background] Momenzadeh S, Koosha A, Kazempoor Monfared M, Bairami J, Zali A, Ommi D, Hosseini B, Hashemi M, Sayadi S, Aryani R, Nematollahi F, Nematollahi L, Barati M. The Effect of Percutaneous Laser Disc Decompression on Reducing Pain and Disability in Patients With Lumbar Disc Herniation. J Lasers Med Sci. 2019 Winter;10(1):29-32. doi: 10.15171/jlms.2019.04. Epub 2018 Dec 15. PMID 31360365
- [Background] Schneider B, Zheng P, Mattie R, Kennedy DJ. Safety of epidural steroid injections. Expert Opin Drug Saf. 2016 Aug;15(8):1031-9. doi: 10.1080/14740338.2016.1184246. Epub 2016 May 13. PMID 27148630
- [Background] Choy DS. Percutaneous laser disc decompression. J Clin Laser Med Surg. 1995 Jun;13(3):125-6. doi: 10.1089/clm.1995.13.125. PMID 10150634
- [Derived] Budrovac D, Rados I, Hnatesen D, Harsanji-Drenjancevic I, Tot OK, Katic F, Lukic I, Skiljic S, Neskovic N, Dimitrijevic I. Effectiveness of Epidural Steroid Injection Depending on Discoradicular Contact: A Prospective Randomized Trial. Int J Environ Res Public Health. 2023 Feb 19;20(4):3672. doi: 10.3390/ijerph20043672. PMID 36834367

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-09-26): https://cdn.clinicaltrials.gov/large-docs/91/NCT05601791/Prot_SAP_ICF_000.pdf